CLINICAL TRIAL: NCT00925223
Title: Study of Brain-derived Neurotrophic Factor in Visceral Hyperalgesia in IBS Patients
Brief Title: Brain-derived Neurotrophic Factor Participates in Visceral Hyperalgesia in Irritable Bowel Syndrome (IBS) Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shandong University (Other)
Responsible Party: Yanqing Li, Qilu hospital of Shandong University
Other Study IDs: 2009SDU-QILU-G02; NSFC30570831
Record Dates: First submitted 2009-06-18; First posted 2009-06-22 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; BDNf; visceral hypersensitivity
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — two mucosal biospecimens will be obtained from the rectosigmoid junction from each patient.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- irritable bowel syndrome: patients with diarrhea-predominant IBS will be enrolled in this group.
- control group: patients with colon cancer or colon polyp will be enrolled as control group.

SUMMARY:
Brain-derived neurotrophic factor (BDNF), originally known to be a member of the nerve growth factor family, has aroused attention as a modulator in visceral hyperalgesia recently. Visceral hypersensitivity is recognized as a clinical hallmark in IBS patients. So in this study, the investigators will focus on the role of BDNF in colonic hyperalgesia in IBS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with irritable bowel syndrome.

Exclusion Criteria:

* Patients have similar clinical symptoms as IBS, yet there is morphologic changes in the intestine.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Irritable bowel syndrome (IBS) is a common functional gastrointestinal disorder characterized by recurrent abdominal pain or discomfort associated with altered bowel habits in the absence of structural and biochemical abnormalities.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-08 (Estimated); Study Completion 2009-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD. MD., Study Director — Department of Gastroenterology, Qilu Hospital, Shandong University